CLINICAL TRIAL: NCT00005287
Title: Late Sequelae of Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2008; R01HL036796 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Lung Diseases; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Lung Diseases; Bronchopulmonary Dysplasia

SUMMARY:
To measure the cardiopulmonary function in individuals who developed bronchopulmonary dysplasia (BPD) at Stanford University Medical Center from 1964-1973 and to determine the factors associated with the presence of cardiopulmonary function abnormalities in these adolescents and young adults.

DETAILED DESCRIPTION:
BACKGROUND:

Eleven to 22 percent of prematurely born human infants with Respiratory Distress Syndrome (RDS) treated with artificial ventilation and supplemental oxygen therapy, develop a severe chronic lung disease called bronchopulmonary dysplasia. While many children who had BPD are asymptomatic by three years of age, some can have respiratory symptoms and abnormal pulmonary function tests at nine years of age. The hypothesis tested in this study is that abnormalities of pulmonary function seen in infants with BPD can persist into adolescence, even in asymptomatic children and young adults.

DESIGN NARRATIVE:

A detailed interval pulmonary history was taken. Pulmonary abnormalities were determined by pulmonary angiography and lateral chest x-ray and pulmonary function tests for small airway obstruction, reversible bronchial hyperreactivity, distribution of ventilation, air trapping and hyperinflation, residual interstitial disease or edema, vascular bed loss, and gas exchange. Right and left ventricular hypertrophy were evaluated by electrocardiogram. Elevated right ventricular pressure was estimated by echocardiography with doppler ultrasound. The atopic status of the children was determined. Other abnormalities, including growth retardation, developmental delay, hearing loss, retrolental fibroplasia, and neurologic disability seen in BPD were assessed by history and physical examination.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-07; Study Completion 1989-06

REFERENCES:
- [Background] Northway WH Jr, Moss RB, Carlisle KB, Parker BR, Popp RL, Pitlick PT, Eichler I, Lamm RL, Brown BW Jr. Late pulmonary sequelae of bronchopulmonary dysplasia. N Engl J Med. 1990 Dec 27;323(26):1793-9. doi: 10.1056/NEJM199012273232603. PMID 2247118